CLINICAL TRIAL: NCT00139230
Title: TPLF-4, Compressed TPLF for Locally Advanced Squamous Cell Carcinoma
Brief Title: Combination Chemotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96-184
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Squamous Cell Carcinoma; Carcinoma of Head/Neck
Keywords: Squamous Cell Carcinoma of Head and Neck; Compressed TPFL; Taxotere; Growth Factor Support
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; Fluorouracil; Leucovorin; Granulocyte Colony-Stimulating Factor; Ciprofloxacin

INTERVENTIONS:
Drug: Taxotere
Drug: Cisplatin
Drug: 5-Fluorouracil
Drug: Leucovorin
Drug: G-CSF
Drug: Ciprofloxacin

SUMMARY:
The purpose of this study is to further test a combination chemotherapy regimen for the treatment of squamous cell carcinoma of the head and neck and to see if the addition of supportive medicine can help reduce the side effects of these drugs.

DETAILED DESCRIPTION:
* Patients will be admitted to hospital and receive a one hour infusion of taxotere. Approximately 2 hours after taxotere is finished they will receive cisplatin, 5-fluorouracil, and leucovorin continuously over a 4 day period.
* Approximately 6-12 hours after the chemotherapy ends patients will be given growth factor support and ciprofloxacin until the patient's ANC level is greater than 10,000.
* Infusion of chemotherapy will be repeated every 28 days (1 cycle is 28 days).
* During each cycle patients will have blood tests performed weekly and may be asked to return to the Head and Neck Clinic for examination around the middle of each cycle.
* At the end of each cycle the impact of the chemotherapy will be assessed. If after 2 cycles, the cancer has not responded sufficiently the patient will not receive any more chemotherapy. However, if significant reduction in the size of the patients tumor is observed, a third and final cycle will be performed.
* During the fourth or fifth week of cycle 3, patients will undergo re-staging evaluation under anesthesia with primary-site biopsies and planning of radiotherapy.
* Within 2 weeks of completion of chemotherapy cycle 3 all patients will receive twice daily radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of squamous cell carcinoma of head and neck.
* All patients with previously untreated Stage III or IV.
* Measurable disease
* Complete recovery from previous diagnostic or therapeutic procedures.
* Life expectancy greater than 3 months
* Creatinine less than or equal to 1.5
* SGOT less than 1.5 x ULN
* Alkaline phosphatase less than 2.5 x ULN
* WBC greater than or equal to 4,000/mm
* Platelet count greater than to equal to 100,000/mm
* Hemoglobin greater than or equal to 10gm/dl
* Patients of childbearing age must use effective contraception methods.

Exclusion Criteria:

* Patients with previous head and neck cancer except those treated with surgery only.
* Patients with concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Peripheral neuropathy exceeding grade 1.
* Cardiovascular or pulmonary disease
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1997-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a four day regimen of taxotere, cisplatin, 5-fluorouracil and high-dose leucovorin with growth factor support and ciprofloxacin.

SECONDARY OUTCOMES:
To determine the efficacy of this regimen in patients with advances, previously untreated squamous cell carcinoma of the head and neck.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Haddad R, Colevas AD, Tishler R, Busse P, Goguen L, Sullivan C, Norris CM, Lake-Willcutt B, Case MA, Costello R, Posner M. Docetaxel, cisplatin, and 5-fluorouracil-based induction chemotherapy in patients with locally advanced squamous cell carcinoma of the head and neck: the Dana Farber Cancer Institute experience. Cancer. 2003 Jan 15;97(2):412-8. doi: 10.1002/cncr.11063. PMID 12518365
- [Background] Colevas AD, Norris CM, Tishler RB, Lamb CC, Fried MP, Goguen LA, Gopal HV, Costello R, Read R, Adak S, Posner MR. Phase I/II trial of outpatient docetaxel, cisplatin, 5-fluorouracil, leucovorin (opTPFL) as induction for squamous cell carcinoma of the head and neck (SCCHN). Am J Clin Oncol. 2002 Apr;25(2):153-9. doi: 10.1097/00000421-200204000-00010. PMID 11943893
- [Background] Goguen LA, Posner MR, Tishler RB, Wirth LJ, Norris CM, Annino DJ, Sullivan CA, Li Y, Haddad RI. Examining the need for neck dissection in the era of chemoradiation therapy for advanced head and neck cancer. Arch Otolaryngol Head Neck Surg. 2006 May;132(5):526-31. doi: 10.1001/archotol.132.5.526. PMID 16702569
- [Background] Haddad R, Tishler R, Wirth L, Norris CM, Goguen L, Sullivan C, O'Donnell L, Li Y, Posner M. Rate of pathologic complete responses to docetaxel, cisplatin, and fluorouracil induction chemotherapy in patients with squamous cell carcinoma of the head and neck. Arch Otolaryngol Head Neck Surg. 2006 Jun;132(6):678-81. doi: 10.1001/archotol.132.6.678. PMID 16785415